CLINICAL TRIAL: NCT03416036
Title: Evaluation of the Efficacy of the Live Attenuated Tetravalent Dengue Vaccine Against DENV-2 and DENV-3 Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 323
Record Dates: First submitted 2018-01-24; First posted 2018-01-30 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: TV003 + rDEN2Δ30-7169 (Experimental): Participants will receive a single dose of TV003 at study entry (Day 0) and rDEN2Δ30-7169 on Day 28.
  Interventions: Biological: TetraVax-DV-TV003 (TV003); Biological: rDEN2Δ30-7169 (DENV-2)
- Arm 2: TV003 + rDEN3Δ30 (Experimental): Participants will receive a single dose of TV003 at study entry (Day 0) and rDEN3Δ30 on Day 28.
  Interventions: Biological: TetraVax-DV-TV003 (TV003); Biological: rDEN3Δ30 (DENV-3)
- Arm 3: Placebo + rDEN2Δ30-7169 (Placebo Comparator): Participants will receive placebo at study entry (Day 0) and rDEN2Δ30-7169 on Day 28.
  Interventions: Biological: rDEN2Δ30-7169 (DENV-2); Biological: Placebo
- Arm 4: Placebo + rDEN3Δ30 (Placebo Comparator): Participants will receive placebo at study entry (Day 0) and rDEN3Δ30 on Day 28.
  Interventions: Biological: rDEN3Δ30 (DENV-3); Biological: Placebo

INTERVENTIONS:
Biological: TetraVax-DV-TV003 (TV003) — TV003 contains 10^3.3 plaque-forming units (PFU)/mL of rDEN1Δ30, 10^3.3 PFU/mL of rDEN2/4Δ30(ME), 10^3.3 PFU/mL of rDEN3Δ30/31-7164, and 10^3.3 PFU/mL of rDEN4Δ30. Administered by subcutaneous injection in the deltoid region of the upper arm
  Arms: Arm 1: TV003 + rDEN2Δ30-7169; Arm 2: TV003 + rDEN3Δ30
Biological: rDEN2Δ30-7169 (DENV-2) — Administered at a dose of 10^3 PFU by subcutaneous injection in the deltoid region of the upper arm
  Arms: Arm 1: TV003 + rDEN2Δ30-7169; Arm 3: Placebo + rDEN2Δ30-7169
Biological: rDEN3Δ30 (DENV-3) — Administered at a dose of 10^3 PFU by subcutaneous injection in the deltoid region of the upper arm
  Arms: Arm 2: TV003 + rDEN3Δ30; Arm 4: Placebo + rDEN3Δ30
Biological: Placebo — Administered by subcutaneous injection in the deltoid region of the upper arm
  Arms: Arm 3: Placebo + rDEN2Δ30-7169; Arm 4: Placebo + rDEN3Δ30

SUMMARY:
The purpose of this study is to evaluate the ability of a single dose of a live attenuated recombinant tetravalent dengue vaccine (TetraVax-DV-TV003, referred to as TV003) to protect against infection with a controlled human infection strain of either DENV-2 (rDEN2Δ30-7169) or DENV-3 (rDEN3Δ30) in adults 18 to 50 years of age with no history of previous flavivirus infection.

DETAILED DESCRIPTION:
This study will evaluate the ability of a single dose of a live attenuated recombinant tetravalent dengue vaccine (TetraVax-DV-TV003, referred to as TV003) to protect against infection with a controlled human infection strain of either DENV-2 (rDEN2Δ30-7169) or DENV-3 (rDEN3Δ30) in adults 18 to 50 years of age with no history of previous flavivirus infection.

Participants will be randomly assigned to receive either TV003 or placebo at study entry (Day 0) and either rDEN2Δ30-7169 or rDEN3Δ30 on Day 28.

Study visits will occur on Days 0, 4, 6, 8, 10, 12, 14, 16, 21, 28, 32, 34, 36, 38, 40, 42, 44, 49, 56, 84, 118, and 208. Visits may include a physical examination and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive.
* Good general health as determined by physical examination, laboratory screening, and review of medical history.
* Available for the duration of the study, which is approximately 28 weeks.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females only: Female subjects of childbearing potential should be willing to use effective contraception and have no plans to undergo IVF (in vitro fertilization) during participation in the trial. Reliable methods of contraception include hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter with a male). All female subjects will be considered as having childbearing potential, except for those who have had a hysterectomy, tubal ligation, or tubal coil (at least 3 months prior to vaccination), or are considered to be post-menopausal, as documented by at least 1 year since last menstrual period.

Exclusion Criteria:

* Females only: Currently pregnant, as determined by positive β-human choriogonadotropin (HCG) test, or breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the requirements of the study protocol.
* Screening laboratory values of Grade 1 or above for absolute neutrophil count (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol.
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by subject history.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* HIV infection, as indicated by screening and confirmatory assays.
* Hepatitis C virus (HCV) infection, as indicated by screening and confirmatory assays.
* Hepatitis B virus (HBV) infection, as indicated by hepatitis B surface antigen (HBsAg) screening.
* Any known immunodeficiency syndrome.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg of a prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or a killed vaccine within 14 days prior to vaccination, or anticipated receipt of any vaccine during the 28 days following vaccination.
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination.
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis Encephalitis virus, or West Nile virus). Subjects will also be screened for Zika virus if they have traveled to areas of South and Central America in the past 18 months that have reported Zika-virus transmission (per the Centers for Disease Control and Prevention Zika travel information).
* Previous receipt of a flavivirus vaccine (licensed or experimental).
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination.
* Definite plans to travel to a dengue-endemic area during the study.
* Refusal to allow specimen storage for future research.

Inclusion Criteria for Challenge with rDEN2Δ30-7169 or rDEN3Δ30

* Currently enrolled in the study.
* Good general health as determined by physical examination and review of medical history.
* Available for the duration of the study, which is approximately 24 weeks after challenge.
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Females only: Female subjects of childbearing potential should be willing to use effective contraception for the duration of the trial. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, and abstinence (greater than or equal to 6 months since last sexual encounter). All female subjects will be considered as having childbearing potential, except for those who have had a hysterectomy, tubal ligation, or tubal coil (at least 3 months prior to vaccination), or who are considered to be post-menopausal, as documented by at least 1 year since last menstrual period.

Exclusion Criteria for rDEN3Δ30 or rDEN2Δ30-7169 Challenge:

* Anaphylaxis or angioedema following TV003 administration.
* Females only: Currently pregnant, as determined by positive β- HCG test, or breast-feeding.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease based on history, physical examination, and/or laboratory studies.
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the subject's ability to understand and cooperate with the requirements of the study protocol.
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, or would render the subject unable to comply with the protocol.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (emergency room visit or hospitalization within the last 6 months).
* Any known immunodeficiency syndrome.
* Current use of anticoagulant medications (this does not include anti-platelet medication such as aspirin or non-steroidal anti-inflammatory medications).
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following challenge. An immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg of a prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine (other than TV003) within 28 days prior to challenge or the anticipated receipt of a live vaccine within 28 days after challenge.
* Receipt of a killed vaccine within 14 days prior to challenge or anticipated receipt of a killed vaccine within 14 days following challenge.
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin, or anticipated receipt of any blood products or immunoglobulin during the 28 days following challenge.
* Anticipated receipt of any other investigational agent in the 28 days before or after challenge.
* Definite plans to travel to a dengue-endemic area during the study.
* Refusal to allow specimen storage for future research.

Other Treatments and Ongoing Exclusion Criteria:

* The following criteria will be reviewed on study day 28 following receipt of TV003 and at study days 28 and 56 following receipt of rDEN2Δ30-7169 or rDEN3Δ30. If any become applicable during the study, the subject will not be included in per-protocol immunogenicity evaluations, as of the exclusionary visit. The subject will, however, be encouraged to remain in the study for safety evaluations until 6 months following the last vaccination (or challenge) received. If the subject had samples obtained at one or more of the protocol-defined time points for immunogenicity, he/she will be included in the intention-to-treat immunogenicity analysis.
* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day post-inoculation period.
* Chronic administration (greater than or equal to 14 days) of steroids (defined as a prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or other immune-modifying drugs initiated during the 28-day period post-inoculation (topical and nasal steroids are allowed).
* Receipt of a licensed killed vaccine during the 14-day post-inoculation period.
* Receipt of immunoglobulins and/or any blood products during the 28-day post-inoculation period.
* Pregnancy (see clarifying language in the protocol) - If the pregnancy is terminated spontaneously or by therapeutic abortion, immunogenicity assessments will be done on blood samples obtained after the pregnancy is terminated.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Frequency of rDEN2Δ30-7160 viremia | Measured through Month 1
  Based on statistical analysis of laboratory evaluations
Frequency of rDEN3Δ30 viremia | Measured through Month 1
  Based on statistical analysis of laboratory evaluations
Occurrence of solicited local and general adverse events (AEs) | Measured through Day 56
  Evaluated using the Adverse Event Grading Table in the study protocol
Occurrence of unsolicited AEs | Measured through Day 56
  Evaluated using the Adverse Event Grading Table in the study protocol
Occurrence of serious adverse events (SAEs) | Measured through Day 208
  Evaluated using the Adverse Event Grading Table in the study protocol

SECONDARY OUTCOMES:
Frequency of viremia after vaccination with TV003 | Measured through Day 208
  Based on statistical analysis of laboratory evaluations
Number of TV003 recipients infected with vaccine virus DENV-1, DENV-2, DENV-3, and DENV-4 | Measured through Day 208
  As defined by recovery of vaccine virus from the blood or serum of a subject and/or seropositivity OR seroconversion to DENV
Serum plaque reduction neutralization titer 50% (PRNT50) to DENV-1, DENV-2, DENV-3, and DENV-4 viruses | Measured through Day 180
  Determined by seropositivity and seroconversion frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Vaccine Testing Center, University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Kirkpatrick BD, Whitehead SS, Pierce KK, Tibery CM, Grier PL, Hynes NA, Larsson CJ, Sabundayo BP, Talaat KR, Janiak A, Carmolli MP, Luke CJ, Diehl SA, Durbin AP. The live attenuated dengue vaccine TV003 elicits complete protection against dengue in a human challenge model. Sci Transl Med. 2016 Mar 16;8(330):330ra36. doi: 10.1126/scitranslmed.aaf1517. Epub 2016 Mar 16. PMID 27089205

DOCUMENTS (1):
  • Informed Consent Form (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT03416036/ICF_000.pdf